CLINICAL TRIAL: NCT05855616
Title: Comparative Study of Two Haemodialysis Catheter Exit Site Dressings: Chlorhexidine Gluconate Dressing vs Chlorhexidine 2% Solution.
Brief Title: Chlorhexidine Dressings for Hemodialysis Catheter Exit Site Care: Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Raquel Pelayo Alonso, Head nurse of the Nephrology department, RN., Hospital Universitario Marqués de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUMV-PIE2020-02
Record Dates: First submitted 2023-02-09; First posted 2023-05-11 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis Catheter Infection

STUDY DESIGN:
Intervention Model Description: Group A: Haemodialysis catheter exit site dressing with 2% chlorhexidine gluconate self-adhesive semi-permeable polyurethane dressings
  Group B: Haemodialysis catheter exit site dressing with 2% chlorhexidine aqueous solution and covered with a dressing of self-adhesive semi-permeable polyurethane dressings.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group "chlorhexidine dressing" (Experimental): CHG Chlorhexidine Gluconate dressing
  Interventions: Device: Group "chlorhexidine dressing"
- Group "solution" (Other): 2% aqueous-based chlorhexidine solution and covering with a semi-permeable self-adhesive polyurethane dressing.
  Interventions: Other: Group "solution"

INTERVENTIONS:
Device: Group "chlorhexidine dressing" — Cleaning of the exit site with physiological saline (0.9%), drying with sterile gauze, application of semi-permeable polyurethane dressing with self-adhesive 2% chlorhexidine gluconate, centring the chlorhexidine gluconate band well over the exit site.
  Arms: Group "chlorhexidine dressing"
Other: Group "solution" — Cleansing of the exit site with physiological saline (0.9%), drying with sterile gauze, disinfection with 2% aqueous-based chlorhexidine solution, environmental drying for 30 seconds and covering with a semi-permeable self-adhesive polyurethane dressing.
  Arms: Group "solution"

SUMMARY:
The objective of this study is to compare the rate of hemodialysis catheter-related infections according to the treatment regimen: chlorhexidine gluconate dressing or chlorhexidine solution.

DETAILED DESCRIPTION:
Introduction: The use of CVC as a vascular access for haemodialysis is associated with increased morbidity and mortality (up to 10 times higher in a patient with a CVC compared to an arteriovenous fistula), contributing to poorer patient outcomes and increased haemodialysis-related costs.

Aim: To compare the rate of catheter-related infections (bacteraemia, exit site infection and tunelitis) between haemodialysis catheter exit site dressing with 2% chlorhexidine gluconate self-adhesive semi-permeable polyurethane dressings (AGCD); and dressing with 2% chlorhexidine solution and covered with self-adhesive semi-permeable polyurethane dressing (PD).

Methods: A randomized clinical trial will be conducted to compare the occurrence of local and systemic infections related to hemodialysis catheter. Two care groups will be formed in which AGCD and PD dressings will be used. In addition, other clinical variables, patient satisfaction and dressing-related skin alterations will also be analyzed.

Scientific relevance: Infectious complications related with hemodialysis catheter have an increased morbidity, mortality and incremented costs.

Key words: hemodialysis, Central Venous Catheters, Bacteremia, exit site infection, tunnel infection, chlorhexidine gluconate dressing.

ELIGIBILITY:
Inclusion Criteria:

* Be included in the haemodialysis programme in our unit.
* Being a carrier of a tunneled central venous catheter as vascular access.
* Remain on haemodialysis treatment for at least 3 months in our unit.
* Consent to participate in the study.

Exclusion Criteria:

* Allergy or hypersensitivity to chlorhexidine or intolerance to polyurethane dressing
* Active catheter-related infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Pelayo Alonso, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanholder R, Canaud B, Fluck R, Jadoul M, Labriola L, Marti-Monros A, Tordoir J, Van Biesen W. Diagnosis, prevention and treatment of haemodialysis catheter-related bloodstream infections (CRBSI): a position statement of European Renal Best Practice (ERBP). NDT Plus. 2010 Jun;3(3):234-246. doi: 10.1093/ndtplus/sfq041. No abstract available. PMID 30792802
- [Background] Wang K, Wang P, Liang X, Lu X, Liu Z. Epidemiology of haemodialysis catheter complications: a survey of 865 dialysis patients from 14 haemodialysis centres in Henan province in China. BMJ Open. 2015 Nov 20;5(11):e007136. doi: 10.1136/bmjopen-2014-007136. PMID 26589425
- [Background] Righetti M, Palmieri N, Bracchi O, Prencipe M, Bruschetta E, Colombo F, Brenna I, Stefani F, Amar K, Scalia A, Conte F. Tegaderm CHG dressing significantly improves catheter-related infection rate in hemodialysis patients. J Vasc Access. 2016 Sep 21;17(5):417-422. doi: 10.5301/jva.5000596. Epub 2016 Aug 1. PMID 27516139
- [Background] Wei L, Li Y, Li X, Bian L, Wen Z, Li M. Chlorhexidine-impregnated dressing for the prophylaxis of central venous catheter-related complications: a systematic review and meta-analysis. BMC Infect Dis. 2019 May 16;19(1):429. doi: 10.1186/s12879-019-4029-9. PMID 31096918

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Started | 26 | 27
Completed | 25 | 25
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group "Solution": Clinical characteristics of the "solution" group
- Group "Chlorhexidine Dressing": Clinical characteristics of the "chlorhexidine dressing" group
- Total: Total of all reporting groups
Arm/Group | Group "Solution" | Group "Chlorhexidine Dressing" | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (13) | 68 (15) | 69 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 25 | 50
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Bacteraemia Rate
Description: presence of fever (body temperature ≥38°C) together with a positive blood culture , with no other source of infection.
Time Frame: 3 months
Population: Patients with tunneled central venous catheter for hemodialysis
Measure: Number; unit: episodes
Groups:
- Control Arm "Group Solution": 2% aqueous-based chlorhexidine solution and covering with a semi-permeable self-adhesive polyurethane dressing.
- Experimental Arm "Chlorhexidine Dressing": Cleaning of the exit site with physiological saline (0.9%), drying with sterile gauze, application of semipermeable polyurethane dressing with self-adhesive 2% chlorhexidine gluconate
Arm/Group | Control Arm "Group Solution" | Experimental Arm "Chlorhexidine Dressing"
Number analyzed (Participants) | 25 | 25
episodes | 2 | 1
Statistical Analysis 1: Comparison: Control Arm "Group Solution" vs Experimental Arm "Chlorhexidine Dressing"; Test type: Other; p = 1.00, t-test, 1 sided; Odds Ratio (OR) = 0.533, 95% CI 2-sided [0.048 to 5.892]

2. Primary Outcome: Exit Site Infection Rate
Description: positive culture of pericatheter smear together with presence of inflammatory signs limited to 2 cm around the cutaneous exit site, without upper extension towards the catheter cuff.
Time Frame: 3 months
Population: patients with tunneled central venous catheters for hemodialysis
Measure: Number; unit: episodes
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Number analyzed (Participants) | 25 | 25
episodes | 2 | 12
Statistical Analysis 1: Comparison: Group "Chlorhexidine Dressing" vs Group "Solution"; Test type: Other; p = 0.013, t-test, 1 sided; Odds Ratio (OR) = 0.176, 95% CI 2-sided [0.039 to 0.790]

3. Primary Outcome: Tunnelitis Rate
Description: occurrence of inflammatory signs extending beyond 2 cm from the cutaneous exit site and into the subcutaneous tract of the catheter (tunnelitis). It may or may not be associated with fever and bacteraemia, and may be accompanied by purulent exudate through the cutaneous exit site.
Time Frame: 3 months
Population: patients with tunneled central venous catheters for hemodialysis
Measure: Number; unit: episodes
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Number analyzed (Participants) | 25 | 25
episodes | 0 | 0

4. Secondary Outcome: Patient Satisfaction Rate
Description: SCALE 18: Degree of perception of positive expectations, of the NOC taxonomy will be used.
  It will be evaluated using a 5-point Likert-type scale where 1- Not at all satisfied, 2- Somewhat satisfied, 3- Moderately satisfied, 4- Very satisfied, 5- Completely satisfied.
Time Frame: 3 months
Population: Patients with tunneled central venous catheter for hemodialysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Number analyzed (Participants) | 25 | 25
Participants
  Not at all satisfied | 0 | 0
  Somewhat satisfied | 0 | 2
  Moderately satisfied | 3 | 1
  Very satisfied | 10 | 5
  Completely satisfied | 12 | 17
Statistical Analysis 1: Comparison: Group "Chlorhexidine Dressing" vs Group "Solution"; Test type: Other; p = 0.137, Chi-squared, Corrected

5. Secondary Outcome: Percentage of Hemodialysis Sessions With Skin Lesions
Description: They will be assessed at each hemodialysis session, using the NOC taxonomy Skin lesions, by means of the SCALE 14: Degree of a negative or adverse condition or response.
  A 5-point Likert-type scale will be used, where 1-Severe, 2-Substantial, 3-Moderate, 4-Leve, 5- None.
Time Frame: 3 months
Population: Hemodialysis sessions performed during the follow-up period are analyzed.
Measure: Number; unit: percentage of sessions
Units Other Than Participants: Hemodialysis sessions
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Number analyzed (Participants) | 25 | 25
Number analyzed (Hemodialysis sessions) | 1004 | 1073
percentage of sessions
  Not Skin Lesions | 99.1 | 99
  Skin Lesions | 0.9 | 1
Statistical Analysis 1: Comparison: Group "Chlorhexidine Dressing" vs Group "Solution"; Test type: Other; p = 0.764, Chi-squared, Corrected

6. Secondary Outcome: Percentage of Hemodialysis Sessions With Dressing-related Skin Erythema Rate
Description: They will be assessed at each hemodialysis session, using the NOC taxonomy Erytema, by means of the SCALE 14: Degree of a negative or adverse condition or response.
  A 5-point Likert-type scale will be used, where 1-Severe, 2-Substantial, 3-Moderate, 4-Leve, 5- None.
Time Frame: 3 months
Population: Hemodialysis sessions performed during the follow-up period are analyzed.
Measure: Number; unit: percentage of sessions
Units Other Than Participants: Hemodialysis sessions
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
Number analyzed (Participants) | 25 | 25
Number analyzed (Hemodialysis sessions) | 1004 | 1073
percentage of sessions
  Not Erythema | 98.2 | 99.2
  Erythema | 1.8 | 0.8
Statistical Analysis 1: Comparison: Group "Chlorhexidine Dressing" vs Group "Solution"; Test type: Other; p = 0.055, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group "Chlorhexidine Dressing" | Group "Solution"
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
The main limitation is the limited follow-up time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT05855616/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT05855616/ICF_001.pdf